CLINICAL TRIAL: NCT03952338
Title: Impact of a Farmers' Market Nutrition Coupon Program on Diet Quality and Psychosocial Well-being Among Low-income Adults: A Randomized Controlled Trial
Brief Title: Impact of BC Farmers' Market Nutrition Coupon Program on Diet Quality and Psychosocial Well-being of Low-income Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); British Columbia Farmers' Market Nutrition Coupon Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB18-0508
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2020-06

CONDITIONS: Diet, Healthy; Health Risk Behaviors
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigators will be blinded to group allocation if participants elect to complete data collection by telephone. Participants cannot be blinded to group assignment but will be blinded to the study objectives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Coupons (Experimental): Participants in the FMNCP group will receive 16 coupon sheets (each sheet contains $21 in coupons) over 10-15 weeks (households with 5-8 individuals will receive 32 coupon sheets) to purchase fruits, vegetables, dairy, meat/poultry/fish, eggs, nuts, and cut herbs at participating BC farmers' markets. To ensure participants receive all 16 coupon sheets, community partners will provide two coupon sheets per household during the first 1-6 weeks of the intervention. Participants in the FMNCP group will also be invited to participate in nutrition skill-building activities (e.g., cooking classes) offered by community partners throughout the intervention period, however participation is not required (this is consistent with the existing FMNCP).
  Interventions: Other: Food coupons; Other: Nutrition skill-building
- Control (No Intervention): No intervention provided. Participants will be eligible to participate in the BC Farmers' Market Nutrition Coupon Program during the next farmers' market season (i.e. one year following the current intervention).

INTERVENTIONS:
Other: Food coupons — Participants will receive 16 coupon sheets (each sheet contains $21 in coupons) over 10-15 weeks (households with 5-8 individuals will receive 32 coupon sheets) to purchase fruits, vegetables, dairy, meat/poultry/fish, eggs, nuts, and cut herbs at participating BC farmers' markets.
  Arms: Nutrition Coupons
Other: Nutrition skill-building — Participants will be invited to participate in nutrition skill-building activities throughout the intervention period. To be consistent with the real-world program, the frequency and types of skill-building activities offered will vary by community partner, and participation is not required.
  Arms: Nutrition Coupons

SUMMARY:
The British Columbia (BC) Farmers' Market Nutrition Coupon Program (FMNCP) provides low-income households with $21/week in coupons to purchase healthy foods at farmers' markets and supportive nutrition skill-building activities. This randomized controlled trial will assess the impact of the BC FMNCP on the overall diet quality (primary outcome), diet quality subscores, mental well-being, sense of community, experiences of food insecurity, risk of malnutrition (secondary outcomes) and subjective social status (exploratory outcome) of low-income adults immediately post-intervention and 16 weeks post-intervention.

DETAILED DESCRIPTION:
Background: The British Columbia (BC) Farmers' Market Nutrition Coupon Program (FMNCP) is a healthy eating initiative funded by the BC Ministry of Health. The program provides low-income households with $21/week in coupons to purchase healthy foods at farmers' markets and supportive nutrition skill-building activities. It is not clear if the BC FMNCP is achieving its aims of improving the diet quality, well-being and health of low-income adults, as its outcomes have not been investigated, and studies of similar programs are limited by weak designs that cannot demonstrate causality. This randomized controlled trial will assess the impact of the FMNCP on the overall diet quality (primary outcome), diet quality subscores, mental well-being, sense of community, experiences of food insecurity, risk of malnutrition (secondary outcomes) and subjective social status (exploratory outcome) of low-income adults immediately post-intervention and 16 weeks post-intervention. A qualitative investigation will also explore mechanisms of action and strategies to maximize positive program impacts.

Methods: Low-income adults (≥ 18 years) from up to 15 rural and urban communities will be randomized to a FMNCP intervention (n=132) or a no-intervention control group (n=132), with a 1:1 allocation ratio. An independent researcher from the Clinical Research Unit at the University of Calgary will generate a blocked randomization sequence that stratifies participants into blocks according to sex (male, female), geographic location (rural, urban), pregnancy (yes, no) and breastfeeding (yes, no). In the existing BC FMNCP, community partners distribute one to two sheets of coupons per week (each sheet contains $21 in coupons) to program participants for a total of 16 sheets. Coupons can be used over 16-20 weeks to purchase fruits, vegetables, dairy, meat/poultry/fish, eggs, nuts, and cut herbs at participating BC farmers' markets. However, to allow sufficient time to recruit participants for this study, community partners will distribute 16 coupon sheets to the FMNCP group over 10-15 weeks (households with 5-8 individuals will receive 32 coupon sheets). To ensure participants receive all 16 coupon sheets, community partners will provide two coupon sheets per household during the first 1-6 weeks of the intervention. Participants in the FMNCP group will also be invited to participate in nutrition skill-building activities (e.g., cooking classes). At baseline (0 weeks), immediately post-intervention (10-15 weeks) and 16 weeks post-intervention (26-31 weeks), participants will access a pilot-tested web-based platform to report sociodemographics, health-related variables, mental well-being, sense of community, experiences of food insecurity, risk of malnutrition and subjective social status. Dietary intake will be assessed via two 24-hour dietary recalls at each time point using the Automated Self-Administered Dietary Assessment Tool for Canada (ASA24-Canada-2018). Diet quality scores will be calculated using the Healthy Eating Index-2015. In addition, immediately post-intervention only, participants will report whether they received FMNCP coupons and attended nutrition skill-building activities (to assess contamination of the control group), how often and how much of their own money was spent at farmers' markets during the intervention period and the types of foods purchased.

Data analysis: Descriptive analyses will be conducted to examine participant characteristics by group at each time point. Characteristics of study completers (i.e., provided data 16-weeks post-intervention) and non-completers will also be compared.

Analyses will be intention-to-treat, in which participants will be analysed within the groups to which they were randomized regardless of adherence (e.g., failure to redeem coupons) or dropout. The analyses will include all participants who provided data at baseline. Repeated measures mixed-effect regression will assess differences in mean HEI-2015 scores, HEI-2015 subscores, mental well-being, sense of community, and subjective social status between the FMNCP and control groups immediately post-intervention and 16-weeks post-intervention. Repeated measures multinomial logistic regression will be used to assess differences in the odds of experiencing household food insecurity and risk of malnutrition for the FMNCP group compared to the control group immediately post-intervention and 16-weeks post-intervention. Statistical models will include intervention group (FMNCP vs control), time from baseline, intervention-by-time interaction, blocking variables (i.e., sex, rural/urban, pregnancy, breastfeeding), baseline values of the outcome, and household size as fixed effects covariates. Participant-specific (i.e., repeated measures) variations in outcomes will be modeled using random effects. Models will also include covariates specific to each outcome to increase the precision of estimates (86). For the primary outcome of overall diet quality, models will include the following: children living in the home (yes, no), sex, age, BMI, marital status, race/ethnicity, perceived health, smoking, day of data collection, and educational level. Adjusted group differences (i.e., FMNCP group vs control group) in outcomes will be estimated using 95% confidence intervals and corresponding p-values.

Subgroup analyses will examine whether the impact of the intervention on primary and secondary outcomes differs according to age group or sex. Dose-response analyses will examine whether the impact of the BC FMNCP on overall diet quality depends on the number of coupons redeemed and the number of nutrition skill-building activities attended. Interactions will be retained in statistical models if p<0.10. Analyses will be conducted in Stata (v15.1, Stata Corp, TX, USA), with p<0.05 indicating statistically significant differences between groups. Data interpretation will jointly consider effect sizes, confidence intervals and statistical significance.

Expected outcomes: Findings will show whether and how a scalable population-level policy that links the agricultural and health sectors influences diet quality, psychosocial well-being and other outcomes among low-income adults. Study findings will inform program adjustments to improve participant outcomes. Other jurisdictions can use these data to determine whether and how to initiate similar programs.

Post-hoc analysis: In a post-hoc analysis, a random forest model will be used to explore heterogeneity of program effects on diet quality (total HEI-2015 scores) among different subgroups of FMNCP study participants. Candidate predictors entered into the algorithm will include all variables examined at baseline, including sociodemographic characteristics (e.g., age, sex, and income) and health-related variables (e.g., self-rated health and smoking). The outcome of the random forest analysis will be total HEI-2015 scores for both the FMNCP and control groups.

ELIGIBILITY:
Individuals will be eligible to participate if they meet the following criteria:

* Adults (age ≥ 18 years)
* Low-income as determined by community-specific thresholds (~$18,000/year annual household income before taxes)
* No expected change in household income prior to study completion (March 2020)
* 8 or fewer people living in the home (including the participant)
* No expected change in household composition prior to study completion (March 2020)
* Primary food shopper for the household
* Does not have self-reported dementia or Alzheimer's Disease
* Able to speak, read and write in English (or have someone who can assist them)
* No plans to move from principal residence prior to study completion (March 2020)
* Has not previously participated in the BC FMNCP

Exclusion Criteria:

• Does not meet one or more inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Olstad, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- Community Partners, Rural and Urban, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aktary ML, Dunn S, Sajobi T, O'Hara H, Leblanc P, McCormack GR, Caron-Roy S, Ball K, Lee YY, Nejatinamini S, Reimer RA, Pan B, Minaker LM, Raine KD, Godley J, Downs S, Nykiforuk CI, Olstad DL. Impact of a farmers' market healthy food subsidy on the diet quality of adults with low incomes in British Columbia, Canada: a pragmatic randomized controlled trial. Am J Clin Nutr. 2023 Apr;117(4):766-776. doi: 10.1016/j.ajcnut.2023.01.017. Epub 2023 Feb 1. PMID 36804420
- [Derived] Aktary ML, Caron-Roy S, Sajobi T, O'Hara H, Leblanc P, Dunn S, McCormack GR, Timmins D, Ball K, Downs S, Minaker LM, Nykiforuk CI, Godley J, Milaney K, Lashewicz B, Fournier B, Elliott C, Raine KD, Prowse RJ, Olstad DL. Impact of a farmers' market nutrition coupon programme on diet quality and psychosocial well-being among low-income adults: protocol for a randomised controlled trial and a longitudinal qualitative investigation. BMJ Open. 2020 May 5;10(5):e035143. doi: 10.1136/bmjopen-2019-035143. PMID 32371514
- See also: BC Farmers' Market Nutrition Coupon Program — https://bcfarmersmarket.org/coupon-program/how-it-works/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community partners recruited study participants throughout BC from June to August 2019 from among their existing clients who were on the FMNCP waitlist in-person or via phone or email. Those who were interested in participating were provided details about the study and screened for eligibility. The first participant was enrolled on June 3, 2019 and the last participant was enrolled on August 23, 2019.
Pre-assignment Details: 285 participants agreed to participate in the study following completion of the informed consent process and were randomized.
Groups:
- FMNCP Group: Study participants in the FMNCP group received 16 coupon sheets valued at CAD $21/sheet over 10-15 weeks to purchase healthy foods from farmers' markets and were eligible to participate in nutrition skill-building activities.
- Control Group: Study participants in the control group did not receive coupons and were not eligible to participate in nutrition skill-building activities.
Period: Overall Study
Arm/Group | FMNCP Group | Control Group
Started | 143 | 142
Completed | 130 | 124
Not Completed | 13 | 18
Not completed — Lost to Follow-up | 11 | 17
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMNCP Group | Control Group | Total
Number analyzed (Participants) | 143 | 142 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (16.0) | 41.5 (16.2) | 42.6 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 128 | 258
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 47 | 50 | 97
  Race/Ethnicity: Black | 3 | 5 | 8
  Race/Ethnicity: East or Southeast Asian | 14 | 11 | 25
  Race/Ethnicity: South or West Asian | 46 | 44 | 90
  Race/Ethnicity: Indigenous | 15 | 10 | 25
  Race/Ethnicity: Other | 4 | 8 | 12
  Race/Ethnicity: Missing | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  Canada | 143 | 142 | 285
Healthy Eating Index 2015 scores [Mean (Standard Deviation); unit: units on a scale] — Diet quality was calculated using the validated Healthy Eating Index-2015 (HEI-2015). HEI-2015 scores reflect adherence to the 2015-2020 Dietary Guidelines for Americans. HEI-2015 scores were calculated by summing component scores for adequacy (total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids) and moderation (refined grains, sodium, added sugars, saturated fats) components. HEI-2015 total scores can range from 0-100, with a higher score indicating a higher diet quality.
  units on a scale | 60.1 (14.3) | 60.4 (14.7) | 60.2 (14.5)
Household food insecurity [Count of Participants; unit: Participants] — Household food insecurity was assessed using a modified version of the Household Food Security Survey Module (HFSSM). The HFSSM was modified to examine experiences of short-term household food insecurity over the past 30 days rather than the past 12 months and response options to questions pertaining to the frequency of experiences (i.e., "How often did this happen?"), were modified to reflect weeks rather than months.
  Participants
    Food secure | 24 | 36 | 60
    Marginal food insecurity | 15 | 9 | 24
    Moderate food insecurity | 57 | 59 | 116
    Severe food insecurity | 38 | 32 | 70
    Missing | 9 | 6 | 15
Malnutrition risk [Count of Participants; unit: Participants] — Malnutrition risk was assessed using the Malnutrition Universal Screening Tool. Population: Participants who were pregnant or breastfeeding (n=39) were excluded given the changes in weight and body composition throughout these life stages.
  Participants
    number analyzed (Participants) | 124 | 124 | 248
    Low | 101 | 94 | 195
    Medium | 14 | 18 | 32
    High | 8 | 11 | 19
    Missing | 1 | 1 | 2
Mental Well-being [Mean (Standard Deviation); unit: units on a scale] — Mental well-being was measured using the Warwick-Edinburgh Mental Well-Being Scale (total possible score 14 to 70).
  units on a scale | 48.1 (10.4) | 49.4 (10.5) | 48.8 (10.5)
Sense of community [Mean (Standard Deviation); unit: units on a scale] — Sense of community was assessed using the 8-item Brief Sense of Community Scale (total possible score 8 to 40).
  units on a scale | 29.6 (5.5) | 29.4 (6.0) | 29.5 (5.8)
Subjective social status [Mean (Standard Deviation); unit: units on a scale] — Subjective social status was measured using the MacArthur Scale of Subjective Social Status community scale (scale from 1 to 10).
  units on a scale | 6.0 (2.1) | 6.0 (2.2) | 6.0 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Intervention and Control Groups in Mean Overall Diet Quality by Healthy Eating Index-2015 Scores Immediately Post-intervention (10-15 Weeks)
Description: Difference between intervention and control groups in mean overall diet quality by Healthy Eating Index-2015 scores immediately post-intervention (10-15 weeks). Healthy Eating Index-2015 scores are calculated from 24-hour dietary recalls and can range from 0-100, with a higher score indicating higher diet quality.
Time Frame: post-intervention (10-15 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 63.6 (1.3) | 62.1 (1.3)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.97, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-4.07 to 3.93]

2. Primary Outcome: Difference Between Intervention and Control Groups in Mean Overall Diet Quality by Healthy Eating Index-2015 Scores at 16 Weeks Post-intervention (26-31 Weeks)
Description: Difference between intervention and control groups in mean overall diet quality by Healthy Eating Index-2015 scores at 16 weeks post-intervention (26-31 weeks). Healthy Eating Index-2015 scores are calculated from 24-hour dietary recalls and can range from 0-100, with a higher score indicating higher diet quality.
Time Frame: 16 weeks post-intervention (26-31 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 62.0 (1.4) | 59.2 (1.4)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.57, Mixed Models Analysis; Mean Difference (Final Values) = 1.22, 95% CI 2-sided [-3.00 to 5.44]

3. Secondary Outcome: Difference Between Intervention and Control Groups in Mean Mental Well-being Scores by Warwick-Edinburgh Mental Well-Being Scale Immediately Post-intervention (10-15 Weeks)
Description: Items on the 14-item Warwick-Edinburgh Mental Well-Being Scale are self-reported over the past two weeks. There are 14 items with 5 response categories (1=none of the time; 5=all of the time), summed to provide a single score ranging from 14-70. A higher score indicates higher perceived mental well-being.
Time Frame: post-intervention (10-15 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 48.8 (0.8) | 48.3 (0.8)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [-0.32 to 4.23]

4. Secondary Outcome: Difference Between Intervention and Control Groups in Mean Mental Well-being Scores by Warwick-Edinburgh Mental Well-Being Scale at 16 Weeks Post-intervention (26-31 Weeks)
Description: as for outcome 3
Time Frame: 16 weeks post-intervention (26-31 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 49.5 (0.9) | 48.8 (0.9)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = 2.10, 95% CI 2-sided [-0.22 to 4.43]

5. Secondary Outcome: Difference Between Intervention and Control Groups in Mean Sense of Community by the Brief Sense of Community Scale Immediately Post-intervention (10-15 Weeks)
Description: Items on the 8-item Brief Sense of Community Scale are self-reported in which each item is scored using a Likert Scale of 1 (strongly disagree) to 5 (strongly agree). Scores can range from 8-40. A higher score indicates a stronger sense of community.
Time Frame: post-intervention (10-15 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 28.8 (0.5) | 27.9 (0.5)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-0.17 to 2.46]

6. Secondary Outcome: Difference Between Intervention and Control Groups in Mean Sense of Community by the Brief Sense of Community Scale at 16 Weeks Post-intervention (26-31 Weeks)
Description: as for outcome 5
Time Frame: 16 weeks post-intervention (26-31 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 29.1 (0.5) | 29.4 (0.5)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.95, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-1.39 to 1.30]

7. Secondary Outcome: Difference Between Intervention and Control Groups in the Odds of Experiencing Household Food Insecurity Immediately Post-intervention (10-15 Weeks)
Description: Difference between intervention and control groups in the odds of experiencing household food insecurity immediately post-intervention (10-15 weeks). Items on the 18-item Household Food Security Survey Module are self-reported in relation to experiences in the past month.
Time Frame: post-intervention (10-15 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
Participants
  Food secure | 46 | 35
  Food insecure | 88 | 87
  Missing | 9 | 20
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.01, Regression, Logistic; Odds Ratio (OR) = 0.21, 95% CI 2-sided [0.06 to 0.70]

8. Secondary Outcome: Difference Between Intervention and Control Groups in the Odds of Experiencing Household Food Insecurity at 16 Weeks Post-intervention (26-31 Weeks)
Description: Difference between intervention and control groups in the odds of experiencing household food insecurity at 16 weeks post-intervention (26-31 weeks). Items on the 18-item Household Food Security Survey Module are self-reported in relation to experiences in the past month.
Time Frame: 16 weeks post-intervention (26-31 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
Participants
  Food secure | 49 | 48
  Food insecure | 74 | 73
  Missing | 20 | 21
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.09 to 0.96]

9. Secondary Outcome: Difference Between Intervention and Control Groups in the Odds of Malnutrition by Malnutrition Universal Screening Tool Immediately Post-intervention (10-15 Weeks)
Description: Items on the Malnutrition Universal Screening Tool are self-reported and based on BMI (scored as 0= >20, 1= 18.5-20, 2 = <18.5) and percent of unplanned weight loss in the past 3-4 months (scored as 0 = <5%, 1 = 5-10%, 2 = >10%). Overall risk of malnutrition will be scored as 0=low risk, 1= medium risk, and >= 2= high risk.
Time Frame: post-intervention (10-15 weeks).
Population: Participants who were pregnant or breastfeeding (n=39) were excluded given the changes in weight and body composition throughout these life stages
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 122 | 124
Participants
  Medium/high malnutrition risk | 26 | 20
  Low malnutrition risk | 87 | 91
  Missing | 9 | 13
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.236, Regression, Logistic; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.27 to 7.23]

10. Secondary Outcome: Difference Between Intervention and Control Groups in the Odds of Malnutrition by Malnutrition Universal Screening Tool at 16 Weeks Post-intervention (26-31 Weeks)
Description: as for outcome 9
Time Frame: 16 weeks post-intervention (26-31 weeks).
Population: Participants who were pregnant or breastfeeding were excluded given the changes in weight and body composition throughout these life stages.
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 123 | 124
Participants
  Medium/high malnutrition risk | 24 | 19
  Low malnutrition risk | 83 | 86
  Missing | 16 | 19
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.220, Regression, Logistic; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.62 to 7.97]

11. Secondary Outcome: Difference Between Intervention and Control Groups in Mean Diet Quality Subscores by Healthy Eating Index-2015 Immediately Post-intervention (10-15 Weeks)
Description: Healthy Eating Index (HEI)-2015 scores are calculated from 24-hour dietary recalls. HEI-2015 total scores can range from 0-100, with a higher score indicating a higher diet quality. HEI-2015 total scores are calculated by summing subscores for adequacy components (total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids) and moderation components (refined grains, sodium, added sugars, saturated fats). Possible subscale scores are as follows:
  Adequacy components (higher score indicates a higher intake):
  Total vegetables (0-5) Greens and beans (0-5) Total fruits (0-5) Whole fruits (0-5) Whole grains (0-10) Dairy (0-10) Total protein foods (0-5) Seafood and plant proteins (0-5) Fatty acids (0-10)
  Moderation components (higher score indicates a lower intake) Sodium (0-10) Refined grains (0-10) Saturated fats (0-10) Added sugars (0-10)
Time Frame: post-intervention (10-15 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale
  Total vegetables | 4.3 (0.1) | 4.1 (0.1)
  Greens and beans | 3.3 (0.2) | 2.9 (0.2)
  Total fruits | 3.4 (0.2) | 3.0 (0.2)
  Whole fruits | 3.6 (0.2) | 3.1 (0.2)
  Whole grains | 4.9 (0.4) | 4.3 (0.3)
  Dairy | 5.7 (0.3) | 6.0 (0.3)
  Total protein | 4.3 (0.1) | 4.2 (0.1)
  Seafood and plant proteins | 3.2 (0.2) | 3.0 (0.2)
  Fatty acids | 6.0 (0.4) | 5.8 (0.4)
  Sodium | 3.2 (0.3) | 3.7 (0.3)
  Refined grains | 6.2 (0.3) | 6.8 (0.3)
  Saturated fats | 6.6 (0.3) | 6.5 (0.3)
  Added sugars | 8.9 (0.2) | 8.7 (0.2)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Total vegetables; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.37 to 0.55]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Greens and beans; Test type: Superiority; p = 0.85, Mixed Models Analysis; Median Difference (Final Values) = -0.07, 95% CI 2-sided [-0.84 to 0.69]
Statistical Analysis 3: Comparison: FMNCP Group vs Control Group; Test type: Superiority — Total fruits; p = 0.29, Mixed Models Analysis; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.29 to 0.98]
Statistical Analysis 4: Comparison: FMNCP Group vs Control Group; Whole fruits; Test type: Superiority; p = 0.07, Mixed Models Analysis; Median Difference (Final Values) = 0.60, 95% CI 2-sided [-0.06 to 1.26]
Statistical Analysis 5: Comparison: FMNCP Group vs Control Group; Whole grains; Test type: Superiority; p = 0.92, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-1.16 to 1.05]
Statistical Analysis 6: Comparison: FMNCP Group vs Control Group; Dairy; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-1.29 to 0.89]
Statistical Analysis 7: Comparison: FMNCP Group vs Control Group; Total protein; Test type: Superiority; p = 0.15, Mixed Models Analysis; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.12 to 0.74]
Statistical Analysis 8: Comparison: FMNCP Group vs Control Group; Seafood and plant proteins; Test type: Superiority; p = 0.92, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.78 to 0.71]
Statistical Analysis 9: Comparison: FMNCP Group vs Control Group; Fatty acids; Test type: Superiority; p = 0.67, Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-1.47 to 0.94]
Statistical Analysis 10: Comparison: FMNCP Group vs Control Group; Sodium; Test type: Superiority; p = 0.61, Mixed Models Analysis; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.45 to 0.84]
Statistical Analysis 11: Comparison: FMNCP Group vs Control Group; Refined grains; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-2.34 to 0.04]
Statistical Analysis 12: Comparison: FMNCP Group vs Control Group; Saturated fats; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.51 to 1.57]
Statistical Analysis 13: Comparison: FMNCP Group vs Control Group; Added sugars; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.56 to 0.92]

12. Secondary Outcome: Difference Between Intervention and Control Groups in Mean Diet Quality Subscores by Healthy Eating Index-2015 at 16 Weeks Post-intervention (26-31 Weeks)
Description: as for outcome 11
Time Frame: 16 weeks post-intervention (26-31 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale
  Total vegetables | 4.2 (0.1) | 4.1 (0.1)
  Greens and beans | 3.4 (0.2) | 3.0 (0.2)
  Total fruits | 2.8 (0.2) | 2.6 (0.2)
  Whole fruits | 3.3 (0.2) | 2.8 (0.2)
  Whole grains | 5.3 (0.4) | 3.9 (0.4)
  Dairy | 6.4 (0.3) | 5.1 (0.3)
  Total protein | 4.2 (0.2) | 4.2 (0.2)
  Seafood and plant proteins | 3.1 (0.2) | 2.9 (0.2)
  Fatty acids | 5.2 (0.4) | 6.0 (0.4)
  Sodium | 2.9 (0.3) | 3.8 (0.3)
  Refined grains | 6.3 (0.4) | 5.7 (0.4)
  Saturated fats | 6.1 (0.3) | 6.4 (0.3)
  Added sugars | 8.8 (0.2) | 8.5 (0.2)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Total vegetables; Test type: Superiority; p = 0.85, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.61 to 0.50]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Greens and beans; Test type: Superiority; p = 0.82, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.88 to 0.70]
Statistical Analysis 3: Comparison: FMNCP Group vs Control Group; Total fruits; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.43 to 0.93]
Statistical Analysis 4: Comparison: FMNCP Group vs Control Group; Whole fruits; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-0.04 to 1.46]
Statistical Analysis 5: Comparison: FMNCP Group vs Control Group; Whole grains; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.63 to 1.84]
Statistical Analysis 6: Comparison: FMNCP Group vs Control Group; Dairy; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [0.31 to 2.62]
Statistical Analysis 7: Comparison: FMNCP Group vs Control Group; Total protein; Test type: Superiority; p = 0.39, Mixed Models Analysis; Median Difference (Final Values) = 0.21, 95% CI 2-sided [-0.27 to 0.69]
Statistical Analysis 8: Comparison: FMNCP Group vs Control Group; Seafood and plant proteins; Test type: Superiority; p = 0.81, Mixed Models Analysis; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.90 to 0.70]
Statistical Analysis 9: Comparison: FMNCP Group vs Control Group; Fatty acids; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-2.57 to -0.04]
Statistical Analysis 10: Comparison: FMNCP Group vs Control Group; Sodium; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.86 to 0.48]
Statistical Analysis 11: Comparison: FMNCP Group vs Control Group; Refined grains; Test type: Superiority; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-1.25 to 1.40]
Statistical Analysis 12: Comparison: FMNCP Group vs Control Group; Saturated fats; Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.98 to 1.13]
Statistical Analysis 13: Comparison: FMNCP Group vs Control Group; Added sugars; Test type: Superiority; p = 0.59, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.55 to 0.97]

13. Secondary Outcome: Difference Between Intervention and Control Groups in the Risk of Experiencing Marginal, Moderate, or Severe Household Food Insecurity Immediately Post-intervention (10-15 Weeks)
Description: Difference between intervention and control groups in the risk of experiencing marginal, moderate, or severe household food insecurity (relative to being food secure) immediately post-intervention (10-15 weeks). Items on the 18-item Household Food Security Survey Module are self-reported in relation to experiences in the past month.
Time Frame: post-intervention (10-15 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
Participants
  Food secure | 46 | 35
  Marginal food insecurity | 25 | 24
  Moderate food insecurity | 39 | 35
  Severe food insecurity | 24 | 28
  Missing | 9 | 20
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.01, Mixed Models Analysis — Marginal food insecurity; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 0.15, 95% CI 2-sided [0.03 to 0.67]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Moderate food insecurity; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 0.56, 95% CI 2-sided [0.17 to 1.82]
Statistical Analysis 3: Comparison: FMNCP Group vs Control Group; Severe food insecurity; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 0.16, 95% CI 2-sided [0.03 to 0.76]

14. Secondary Outcome: Difference Between Intervention and Control Groups in the Risk of Experiencing Marginal, Moderate, or Severe Household Food Insecurity at 16 Weeks Post-intervention (26-31 Weeks)
Description: Difference between intervention and control groups in the risk of experiencing marginal, moderate, or severe household food insecurity (relative to being food secure) at 16 weeks post-intervention (26-31 weeks). Items on the 18-item Household Food Security Survey Module are self-reported in relation to experiences in the past month.
Time Frame: 16 weeks post-intervention (26-31 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
Participants
  Food secure | 49 | 48
  Marginal food insecurity | 19 | 14
  Moderate food insecurity | 38 | 31
  Severe food insecurity | 17 | 28
  Missing | 20 | 21
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Marginal food insecurity; Test type: Superiority; p = 0.10, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio, log = 0.28, 95% CI 2-sided [0.06 to 1.29]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Moderate food insecurity; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.21 to 2.21]
Statistical Analysis 3: Comparison: FMNCP Group vs Control Group; Severe food insecurity; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 0.11, 95% CI 2-sided [0.02 to 0.56]

15. Secondary Outcome: Difference Between Intervention and Control Groups in the Risk of Being at a Medium or High Risk of Malnutrition by Malnutrition Universal Screening Tool Immediately Post-intervention (10-15 Weeks)
Description: Difference between intervention and control groups in the risk of being at a medium or high risk of malnutrition (relative to being at low risk of malnutrition) by Malnutrition Universal Screening Tool immediately post-intervention (10-15 weeks). Items on the Malnutrition Universal Screening Tool are self-reported and based on BMI (scored as 0= >20, 1= 18.5-20, 2 = <18.5) and percent of unplanned weight loss in the past 3-4 months (scored as 0 = <5%, 1 = 5-10%, 2 = >10%). Overall risk of malnutrition was scored as 0=low risk, 1= medium risk, and >= 2= high risk.
Time Frame: post-intervention (10-15 weeks).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 122 | 124
Participants
  Low malnutrition risk | 87 | 91
  Medium malnutrition risk | 18 | 9
  High malnutrition risk | 8 | 11
  Missing | 9 | 13
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Medium malnutrition risk; Test type: Superiority; p = 0.15, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 2.94, 95% CI 2-sided [0.68 to 12.66]
Statistical Analysis 2: Comparison: FMNCP Group; High malnutrition risk; Test type: Superiority; p = 0.86, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.20 to 7.13]

16. Secondary Outcome: Difference Between Intervention and Control Groups in the Risk of Being at a Medium or High Risk of Malnutrition by Malnutrition Universal Screening Tool at 16 Weeks Post-intervention (26-31 Weeks)
Description: Difference between intervention and control groups in the risk of being at a medium or high risk of malnutrition (relative to being at low risk of malnutrition) by Malnutrition Universal Screening Tool at 16 weeks post-intervention (26-31 weeks). Items on the Malnutrition Universal Screening Tool are self-reported and based on BMI (scored as 0= >20, 1= 18.5-20, 2 = <18.5) and percent of unplanned weight loss in the past 3-4 months (scored as 0 = <5%, 1 = 5-10%, 2 = >10%). Overall risk of malnutrition was scored as 0=low risk, 1= medium risk, and >= 2= high risk.
Time Frame: 16 weeks post-intervention (26-31 weeks).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 123 | 124
Participants
  Low malnutrition risk | 83 | 86
  Medium malnutrition risk | 14 | 14
  High malnutrition risk | 10 | 5
  Missing | 16 | 19
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Medium malnutrition risk; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.31 to 5.38]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; High malnutrition risk; Test type: Superiority; p = 0.10, Mixed Models Analysis; Mixed effects multinomial logistic regression; Risk Ratio (RR) = 5.48, 95% CI 2-sided [0.73 to 41.3]

17. Other Pre Specified Outcome: Difference Between Intervention and Control Groups in Mean Subjective Social Status by the MacArthur Scale of Subjective Social Status Community Ladder Immediately Post-intervention (10-15 Weeks)
Description: The MacArthur Scale of Subjective Social Status community ladder consists of a self-reported visual analog scale, whereby respondents place themselves on a ladder rung according to their perceived social standing relative to others in their community. Responses can take a value from 1-10, with a higher score indicating higher perceived social status in relation to others' within ones' community.
Time Frame: post-intervention (10-15 weeks).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 5.7 (0.2) | 5.7 (0.2)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.65 to 0.40]

18. Other Pre Specified Outcome: Difference Between Intervention and Control Groups in Mean Subjective Social Status by the MacArthur Scale of Subjective Social Status Community Ladder at 16 Weeks Post-intervention (26-31 Weeks)
Description: as for outcome 17
Time Frame: 16 weeks post-intervention (26-31 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale | 5.9 (0.2) | 5.8 (0.2)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.90, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.57 to 0.50]

19. Other Pre Specified Outcome: Subgroup Analysis for Impact of Intervention on Overall Diet Quality (Assessed by Healthy Eating Index-2015) by Sex Immediately Post-intervention (10-15 Weeks)
Description: Subgroup analysis for impact of intervention on overall diet quality (assessed by Healthy Eating Index-2015) by self-reported sex immediately post-intervention (10-15 weeks). Healthy Eating Index (HEI)-2015 scores are calculated from 24-hour dietary recalls. HEI-2015 total scores can range from 0-100, with a higher score indicating a higher diet quality. HEI-2015 total scores are calculated by summing subscores for adequacy components (total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids) and moderation components (refined grains, sodium, added sugars, saturated fats). Adequacy and moderation components are each scored from 0-5, except for whole grains, dairy, and fatty acids, which are each scored from 0-10. For adequacy components, a higher score indicates a higher intake, whereas, for moderation components, a higher score indicates a lower intake.
Time Frame: post-intervention (10-15 weeks)
Population: Subgroup analysis for impact of intervention on overall diet quality (assessed by Healthy Eating Index-2015) by self-reported sex.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale
  Males: number analyzed (Participants) | 13 | 14
  Males | 58.8 (11.7) | 62.1 (12.9)
  Females: number analyzed (Participants) | 130 | 128
  Females | 62.2 (15.2) | 62.8 (14.8)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.43, Mixed Models Analysis — Males; Mean Difference (Final Values) = -4.07, 95% CI 2-sided [-14.05 to 5.92]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Females; Test type: Superiority; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-3.75 to 4.66]

20. Other Pre Specified Outcome: Subgroup Analysis for Impact of Intervention on Overall Diet Quality (Assessed by Healthy Eating Index-2015) by Age Immediately Post-intervention (10-15 Weeks)
Description: Subgroup analysis for impact of intervention on overall diet quality (assessed by Healthy Eating Index-2015) by self-reported age immediately post-intervention (10-15 weeks). Healthy Eating Index (HEI)-2015 scores are calculated from 24-hour dietary recalls. HEI-2015 total scores can range from 0-100, with a higher score indicating a higher diet quality. HEI-2015 total scores are calculated by summing subscores for adequacy components (total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids) and moderation components (refined grains, sodium, added sugars, saturated fats). Adequacy and moderation components are each scored from 0-5, except for whole grains, dairy, and fatty acids, which are each scored from 0-10. For adequacy components, a higher score indicates a higher intake, whereas, for moderation components, a higher score indicates a lower intake.
Time Frame: post-intervention (10-15 weeks)
Population: Subgroup analysis for impact of intervention on overall diet quality (assessed by Healthy Eating Index-2015) by self-reported age.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale
  Age 18-59 years: number analyzed (Participants) | 112 | 115
  Age 18-59 years | 61.6 (15.4) | 62.0 (15.0)
  Age 60+ years: number analyzed (Participants) | 31 | 27
  Age 60+ years | 62.9 (13.5) | 65.3 (12.9)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Test type: Superiority; p = 0.66, Mixed Models Analysis — Age 18-59 years; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-5.65 to 3.57]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Age 60+ years; Test type: Superiority; p = 0.40, Mixed Models Analysis; Mean Difference (Final Values) = 3.28, 95% CI 2-sided [-4.36 to 10.93]

21. Other Pre Specified Outcome: Subgroup Analysis for Impact of Intervention on Overall Diet Quality (Assessed by Healthy Eating Index-2015) by Sex at 16 Weeks Post-intervention (26-31 Weeks)
Description: Subgroup analysis for impact of intervention on overall diet quality (assessed by Healthy Eating Index-2015) by self-reported sex at 16 weeks post-intervention (26-31 weeks). Healthy Eating Index-2015 scores are calculated from 24-hour dietary recalls.
Time Frame: 16 weeks post-intervention (26-31 weeks)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale
  Males: number analyzed (Participants) | 13 | 14
  Males | 59.1 (11.5) | 59.7 (13.7)
  Females: number analyzed (Participants) | 130 | 128
  Females | 59.9 (15.0) | 60.3 (14.9)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; Males; Test type: Superiority; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = 6.25, 95% CI 2-sided [-9.13 to 21.63]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; Females; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-3.23 to 5.41]

22. Other Pre Specified Outcome: Subgroup Analysis for Impact of Intervention on Overall Diet Quality (Assessed by Healthy Eating Index-2015) by Age at 16 Weeks Post-intervention (26-31 Weeks)
Description: Subgroup analysis for impact of intervention on overall diet quality (assessed by Healthy Eating Index-2015) by self-reported age at 16 weeks post-intervention (26-31 weeks). Healthy Eating Index-2015 scores are calculated from 24-hour dietary recalls.
Time Frame: 16 weeks post-intervention (26-31 weeks)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
score on a scale
  18-59 years: number analyzed (Participants) | 112 | 115
  18-59 years | 59.3 (15.2) | 59.6 (14.9)
  60+ years: number analyzed (Participants) | 31 | 27
  60+ years | 61.5 (12.8) | 62.7 (13.9)
Statistical Analysis 1: Comparison: FMNCP Group vs Control Group; 18-59 years; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-4.76 to 4.66]
Statistical Analysis 2: Comparison: FMNCP Group vs Control Group; 60+ years; Test type: Superiority; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = 3.66, 95% CI 2-sided [-5.48 to 12.80]

23. Other Pre Specified Outcome: Frequency of Purchasing Food in Farmers' Markets
Description: Self-reported frequency of purchasing food in farmers' markets. "How often did you buy food at a farmers' market (using coupons or money)?"
Time Frame: post-intervention (10-15 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
Participants
  Never | 5 | 60
  Less than once per month | 6 | 11
  Once or twice per month | 38 | 27
  One per week | 76 | 18
  More than once per week | 9 | 4
  Missing | 9 | 22

24. Other Pre Specified Outcome: Frequency of Money Spent at Farmers' Markets at Post-intervention (Excluding Coupons)
Description: Self-reported frequency of money spent at farmers' markets (excluding coupons) among participants who reported purchasing foods from farmers' markets. "How often did you spend household money at a farmers' market? Do not include items you bought with coupons (if applicable)."
Time Frame: post-intervention (10-15 weeks)
Population: Includes only participants who reported purchasing foods from farmers' markets
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 129 | 60
Participants
  Never | 43 | 6
  Less than once per month | 21 | 12
  Once or twice per month | 36 | 22
  One per week | 23 | 15
  More than once per week | 4 | 4
  Missing | 2 | 1

25. Other Pre Specified Outcome: Amount of Money Spent at Farmers' Markets
Description: Self-reported amount of money spent at farmers' markets using coupons and own money
Time Frame: post-intervention (10-15 weeks)
Population: Includes only participants who reported spending money at farmers' markets.
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 84 | 53
Participants
  $1 - $5 | 17 | 2
  $6 - $10 | 25 | 9
  $11 - $19 | 26 | 25
  $20 or more | 14 | 14
  Missing | 2 | 3

26. Other Pre Specified Outcome: Objective Data (From Coupons) on Foods Purchased Using Coupons at Farmers' Markets
Description: Number of coupons redeemed to purchase vegetables, fruit, meat and fish, eggs, dairy, cut herbs, and nuts.
Time Frame: Assessed at post-intervention (10-15 weeks)
Measure: Number; unit: Coupons
Units Other Than Participants: Coupons redeemed
Arm/Group | FMNCP Group
Number analyzed (Participants) | 143
Number analyzed (Coupons redeemed) | 12106
Coupons
  Vegetables | 4718
  Fruits | 2125
  Meat and fish | 1348
  Eggs | 1225
  Dairy | 452
  Cut herbs | 57
  Nuts | 2
  Unmarked coupons | 2179

27. Other Pre Specified Outcome: Foods Purchased at Farmers' Markets Using Own Money (Excluding Coupons)
Description: Self-Reported Foods Purchased at Farmers' Markets using own money (excluding coupons).
Time Frame: Assessed at post-intervention (10-15 weeks)
Population: Includes only participants who reported purchasing foods from farmers' markets
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 82 | 53
Participants
  Vegetables | 28 | 31
  Fruits | 12 | 9
  Meat | 13 | 3
  Dairy | 4 | 3
  Eggs | 4 | 1
  Cut herbs | 1 | 0
  Nuts | 0 | 0
  Other | 20 | 6

28. Other Pre Specified Outcome: Nutrition Skill-building Activity Attendance
Description: Self-reported data on attendance to nutrition skill-building activities ("Did you go to nutrition skill building activities offered by your community partner?")
Time Frame: Assessed at post-intervention (10-15 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | FMNCP Group | Control Group
Number analyzed (Participants) | 143 | 142
Participants
  Yes | 45 | 29
  No | 81 | 90
  Missing | 17 | 23

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assessed.
Arm/Group | FMNCP Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Dietary intake data were self-reported and may be affected by misreporting; Data were obtained only from the primary food shopper in the household; Insufficient data to examine participant-specific coupon distribution and redemption; This study was powered to detect a change in diet quality (the primary outcome) and may have been underpowered to detect changes in the secondary and exploratory outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT03952338/Prot_SAP_000.pdf